CLINICAL TRIAL: NCT00166764
Title: A Study on Evaluation of Mental Health Index of Patients With Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700816
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-09

CONDITIONS: Psychiatric Disorders
Keywords: Psychiatric Disorders; Evaluation of Mental Health Index
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Psychiatric patients under the mental impaired influences, their living function were disabled, and their social lives were handicapped consequently. Idea psychiatric treatment is to control the psychiatric symptoms in a better way, to develop efficient psychiatric adjustment, to manage living stress into a lower level, to gradually develop the meaning and value of the patients' lives, and to obtain the satisfaction and happiness in life for them. In order to investigate the satisfaction for psychiatric patients under the current treatment and to evaluate their psychiatric health, it is necessary to measure the mental health status for the psychiatric patients, and to ensure the ideological status of psychiatric treatment. If there is a mental health measurement for the psychiatric patients, we may precisely identify the mental health levels of the patients and their mental disturbances degrees. Accordingly, we may develop efficient procedure to manage the mental health for the psychiatric patients, and to achieve the goal for the idea psychiatric treatment.

In this study, we established the mental health assessment data sheet according to the clinical experiences. It includes mental health index data sheet, mental-and-physical stress response data sheet, mental sustentation data sheet, and supplemented with a general living satisfaction assessment data sheet. We will evaluate the reliability and validity of this study to ensure the usability of these data sheet in clinics. We will also recruit the continuous treated and mentally stabilized patients as subjects. After obtaining their written informed consents, we will go through these mental health assessments to discover the mental health status of these psychiatric patients, and use it as a reference to develop idea psychiatric treatment. We will use ICC test for the repeated measurement validity, Pearson r correlation coefficient within our data analyses to evaluate the validity of the same measurement, and independent t-test to assess the differences between the patient group and the society group (from previously established data files). This study result may evaluate the possible deficits existing in the traditional psychiatric treatment and may be used as a reference for the development of idea psychiatric medicine.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric Disorders

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan Univeristy
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan